CLINICAL TRIAL: NCT05718726
Title: Overwhelming Post-Splenectomy Infections (OPSI) After Cytoreductive Surgery and Hyperthemic Intraperitoneal Chemotherapy: a Prospective Observational Study
Brief Title: Post Splenectomy Infections After Surgery for Peritoneal Malignancies (OPSI)
Acronym: OPSI
Status: Recruiting | Type: Observational
Sponsor: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SPON-BM-1220
Record Dates: First submitted 2021-09-30; First posted 2023-02-08 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Infection;Post Surg Procedure; Peritoneal Cancer
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire, interview or observation study — Questionnaire administered by telephone

SUMMARY:
The spleen is involved in maintaining immunity and plays an important role in the elimination of encapsulated bacteria and parasites. Patients who undergo splenectomy in conjunction with complete CRS for peritoneal malignancy are at risk of overwhelming post-splenectomy infections post-operatively. These patients are therefore administered vaccinations to lower the risk of infections but as they do not completely eliminate the risk, patients are also prescribed prophylactic antibiotics without clear evidence that they are useful in preventing OPSI. The use of prophylactic antibiotics is not without risk with potential short and long-term risks including resistance, interaction with other medication, clostridium difficile infections, fungal infections, other changes to the microbiome and cost. This study will investigate the incidence of OPSI post splenectomy and assess compliance with prophylactic antibiotics. This is an observational study where consented patients will be telephoned at fixed time points which are 1,6,12 weekly and 6 monthly for a period of five years post-operatively. As part of routine care patients will be telephoned by the clinical nurse specialist at weeks 1,6 and 12. In addition to this the research nurse will telephone the patient 6 monthly for a period of 5 years and complete a questionnaire. The research nurse will complete the questionnaire during each telephone call and this should not take more than 20 minutes. At the start of the telephone call, consent will be confirmed each time and the research nurse will check that the patient is still happy to participate before going ahead.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged >18 and <80 years Patients capable of providing informed consent Patients who have a splenectomy in conjunction with complete cytoreductive surgery (CRS) for any pathology

Exclusion Criteria:

- Patients who are <18 and >80 Patients who do not provide informed consent Patients on immunosuppression therapy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the Peritoneal Malignancy Institute, Hampshire Hospitals Foundation Trust, who have had a splenectomy in conjunction with CRS for any pathology.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-03-25 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2031-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of post-splenectomy infections after surgery | Period of 5 years
  Self-reported measure

SECONDARY OUTCOMES:
Compliance with prophylactic antibiotic regime post splenectomy as per national guidelines | Period of 5 years
  Self-reported measure

CONTACTS AND LOCATIONS:
Overall Officials: Brendon Moran, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- The Peritoneal Malignancy Institute, Hampshire Hospitals NHS Foundation Trust, Basingstoke, Hampshire, United Kingdom